CLINICAL TRIAL: NCT06353464
Title: A Translational Understanding of Obesity-Related Phenotypes Using Brain Imaging and Manipulation
Acronym: OPBIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2306009984
Record Dates: First submitted 2024-02-15; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Water

STUDY DESIGN:
Intervention Model Description: individuals consume two distinct preloads at separate sessions
Masking Description: Participants consume two preloads one at each visit, but are not informed which preload is being consumed on which test visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preloads (Experimental): Delivery of two different preloads to all participants, each preload tested on a separate day/participant, prior to consumption of pizza
  Interventions: Other: Ensure and Water

INTERVENTIONS:
Other: Ensure and Water — Ensure, a liquid meal with 9 grams of protein in 8 ounces consumed 20 minutes before eating pizza; and water, 8 ounces consumed 20 minutes before eating pizza

SUMMARY:
This study will examine a potential relationship between family history of obesity, that is whether people with at least one parent who had obesity in adulthood compared to people with two parents who did not have obesity in adulthood, and the ability of protein intake to curb further intake of food.

DETAILED DESCRIPTION:
1) Abstract of the study A positive energy balance (greater intake than expenditure) can explain weight gain and, when protracted, leads to overweight and obesity. The major question addressed in this proposal is if the timing of activation of specific regions of the brain is predictive of excessive food intake. Functional near infra-red spectroscopy (fNIR), seldom used in human eating studies, provides data similar to functional magnetic resonance imaging (fMRI) but allows for measurement of brain activation during food consumption. The investigator's pilot fNIR data reveal that varying patterns of regional PFC activation are associated with "loss of control" over eating, and that only 60% of individuals respond to acute protein intake with a reduction in food intake. Using fNIR and an acute protein challenge, the investigator will assess the effect of family history of obesity in humans on the satiation response to protein and concomitant activation of the prefrontal cortex (PFC). It is hypothesized that activation of the human medial PFC before the lateral PFC will result in greater intake of palatable food in those subjects with a proneness to obesity, and that these subjects will be less sensitive to the satiety-inducing effects of a protein preload. These results should provide an innovative and useful method for assessing risk for developing obesity and usefulness of preventative interventions.

ELIGIBILITY:
Inclusion Criteria

* BMI 20-40
* weight stable for at least 3 months
* no parents with history of obesity in adulthood, or at least one parent with history of obesity in adulthood

Exclusion Criteria

* no current diagnosis of psychiatric disorders
* no current diagnosis of neurological disorders
* no current diagnosis or history of anorexia nervosa
* no current diagnosis or history of bulimia nervosa
* no pregnancy within the last 9 months
* not currently breastfeeding
* no use of investigational medication in the past 6 months
* no use of prescription anti-seizure medications.
* no use of prescription antidepressant medications
* no use of prescription antipsychotic medications

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Grams of pizza consumed | 3-15 minutes
  Ad libitum during the pizza eating episode
Baseline medial prefrontal cortex oxygenated hemoglobin | 20 minutes
  Micromoles per millimeter of oxygenated hemoglobin of the medial prefrontal cortex prior to pizza consumption
Baseline lateral prefrontal cortex oxygenated hemoglobin | 20 minutes
  Micromoles per millimeter of oxygenated hemoglobin of the lateral prefrontal cortex prior to pizza consumption
medial prefrontal cortex Oxygenated hemoglobin concentration | 3-15 minutes
  Micromoles per millimeter of oxygenated hemoglobin of the medial prefrontal cortex during pizza consumption phase
lateral prefrontal cortex Oxygenated hemoglobin concentration | 3-15 minutes
  Micromoles per millimeter of oxygenated hemoglobin of the lateral prefrontal cortex during pizza consumption phase

SECONDARY OUTCOMES:
medial prefrontal cortex Time to Peak Light Intensity | 3-15 minutes
  The time in seconds that it takes for the oxygenated hemoglobin signal to reach peak in the medial prefrontal cortex during the ad libitum eating episode for each preload
lateral prefrontal cortex Time to Peak Light Intensity | 3-15 minutes
  The time in seconds that it takes for the oxygenated hemoglobin signal to reach peak in the lateral prefrontal cortex during the ad libitum eating episode for each preload
Preload Oxygenated Hemoglobin Difference | 5 minutes
  The difference between the oxygenated hemoglobin concentrations obtained under the two different preloads

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No